CLINICAL TRIAL: NCT04381000
Title: The Impact of Quarantine and the Effectiveness of Telerehabilitation in Patients With Chronic Pain During COVID-19 Pandemic.
Brief Title: Quarantine and Telerehabilitation in Chronic Pain Patients During COVID-19 Pandemic.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3
Record Dates: First submitted 2020-05-07; First posted 2020-05-08 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Chronic Pain
Keywords: COVID-19; Quarantine; Musculoskeletal; Telerehabilitation; Psychosocial; Sleep; Exercise
MeSH Terms: conditions — Chronic Pain; COVID-19; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group will not participate in any exercise program.
- Intervention (Experimental): The intervention group will participate in an exercise program for 6 weeks/ 2 sessions per week, for a total of 12 sessions of 30-45 minutes each.
  Interventions: Other: Exercise Group

INTERVENTIONS:
Other: Exercise Group — The group follows warm up exercise (maximum 10 minutes). This consisted of combined, breathing techniques, low-impact aerobic exercises, free range of motion exercises of upper and lower limbs and spine, and coordination-based exercises of hands and feet. Breathing techniques take regular activities such as sitting, walking, and lying down. At the end of this phase, active stretching exercises of major muscles of arm, leg and trunk were performed.
  Arms: Intervention

SUMMARY:
The quarantine during COVID-19 pandemic has changed daily routine. Staying at home for prolonged periods of time can pose a significant challenge for patients with chronic pain. The purpose of the current study is to investigate how the quarantine effects of psychosocial factors, quality of life, sleep, nutrition and physical activity in patients with chronic musculoskeletal pain. Another purpose is to examine whether a telerehabilitation exercise program is effective during the lockdown period.

DETAILED DESCRIPTION:
Participants, both male and female, with chronic musculoskeletal pain for at least 3 months will be included in the study. They will complete some questions about anxiety, depression, sleep, nutrition, quality of life, pain behavior and characteristics, illness perceptions, functioning and daily routine. Questionnaires will be completed twice (first and last week of quarantine, 40 days of duration). A group of patients will follow an exercise program during this time. It will be evaluated the link between the question of physical and psychological factors in the experience of pain in quarantine situation and, also, it will examine whether a telerehabilitation exercise program is effective during the lockdown period.

ELIGIBILITY:
Inclusion Criteria:

* Patient with chronic musculoskeletal pain (Chronic pain will be defined as pain lasting for 3 or more months. Also, pain intensity will be at least 3 on a 0-10 numerical pain rating scale on most days of the last 3 months).
* Patient with sufficient understanding of the Greek language

Exclusion Criteria:

* Patients without being at quarantine
* Systemic diseases such as rheumatoid arthritis, fibromyalgia and/or polymyalgia rheumatic
* Osteoporosis, haemophilia and/or cancer
* Recent surgery or trauma
* Being pregnant or given birth in the preceding year
* Cognitive impairment
* Inability to provide informed consent and/or complete written questionnaires

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Anxiety and Depression | Change From Baseline in HADS at 40 days
  To measure the levels of anxiety and depression Hospital Anxiety and Depression Scale (HADS), will be used. Patients have to score 14 opinions. Seven of the items relate to anxiety and seven relate to depression. A cut-off point of 8/21 for anxiety or depression has been recommended.
Quality of Life and overall health | Change From Baseline in EQ-5D-3L at 40 days
  To measure quality of life, EQ-5D-3L will be used. The EQ-5D-3L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Pain Intensity | Change From Baseline in NPRS Scores at 40 days
  The Numeric Pain Rating Scale (NPRS) is a unidimensional measure of pain intensity in adults and it will be used in the current study. The most commonly used is the 11-item NPRS. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").The NPRS is a valid and reliable scale to measure pain intensity. In this study, will rate current pain intensity and mean pain intensity during the past 7 days.

SECONDARY OUTCOMES:
Quality and patterns of sleep | Change From Baseline in PSQI Scores at 40 days
  The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep in the older adult. PSQI will be used to assess quality and patterns of sleep in the current study. PSQI differentiates "poor" from "good" sleep by measuring seven domains: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction over the last month. The client self-rates each of these seven areas of sleep. Scoring of the answers is based on a 0 to 3 scale, whereby 3 reflects the negative extreme on the Likert Scale. A global sum of "5" or greater indicates a "poor" sleeper. Although there are several questions that request the evaluation of the client's bed mate or roommate, these are not scored, nor reflected in the attached instrument. An update to the scoring: if 5 is not complete or the value is missing, it now counts as a "0".
Patients' illness perceptions | Change From Baseline in BIPQ Scores at 40 days
  Patients' illness perceptions will be measured based on the Brief Illness Perception Questionnaire (BIPQ). The patient has to rate 8 statements on a 10-point scale (1-10). The higher the score, the greater is the extent to which the patient's illness perceptions are threatening him or her.
Disability | Change From Baseline in ODI Scores at 40 days
  Disability will be assessed using Oswestry Disability Index (ODI) that present ten sections cover Pain, Personal Care, Lifting, Walking, Sitting, Standing, Sleeping, Sex Life, Social Life, and Traveling. Each section has six statements reflecting an increasing level of disability. Respondents choose the statement that most applies to them in each section. The first statement is scored 0; the second is scored 1 and so on to 5 for the last statement. The sum of the section scores is divided by 50 if all sections are completed and multiplied by 100 for the final percentage score.

CONTACTS AND LOCATIONS:
Overall Officials: Eleni V Kapreli, MSc,PhD, Study Chair — Clinical Exercise Physiology & Rehabilitation Laboratory,University of Thessaly; Georgios Tsatsakos, PhD, Principal Investigator — TherapyLab
Locations (1):
- Clinical Exercise Physiology and Rehabilitation Laboratory, Lamia, Central Greece, Greece

REFERENCES:
- [Background] Hawryluck L, Gold WL, Robinson S, Pogorski S, Galea S, Styra R. SARS control and psychological effects of quarantine, Toronto, Canada. Emerg Infect Dis. 2004 Jul;10(7):1206-12. doi: 10.3201/eid1007.030703. PMID 15324539
- [Background] Chatterjee K, Chauhan VS. Epidemics, quarantine and mental health. Med J Armed Forces India. 2020 Apr;76(2):125-127. doi: 10.1016/j.mjafi.2020.03.017. Epub 2020 Apr 22. No abstract available. PMID 32327877
- [Background] Torales J, O'Higgins M, Castaldelli-Maia JM, Ventriglio A. The outbreak of COVID-19 coronavirus and its impact on global mental health. Int J Soc Psychiatry. 2020 Jun;66(4):317-320. doi: 10.1177/0020764020915212. Epub 2020 Mar 31. PMID 32233719